CLINICAL TRIAL: NCT04638426
Title: For 12 Weeks, the Multi Center, Randomized, Double Blinded, Placebo Controlled, Parallel, Dose-finding Clinical Study for the Therapeutic Exploration of Safety and Efficacy Assessment of HL237 Tablet in Patients With Rheumatoid Arthritis (Phase IIa)
Brief Title: Phase 2a Clinical Trial of HL237 for Rheumatoid Arthritis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Hanlim Pharm. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HL237-201
Record Dates: First submitted 2020-11-13; First posted 2020-11-20 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Treatment A (Experimental): HL237 tab. 200mg/day
  Interventions: Drug: HL237 tablet
- Treatment B (Experimental): HL237 tab. 400mg/day
  Interventions: Drug: HL237 tablet
- Treatment C (Experimental): HL237 tab. 800mg/day
  Interventions: Drug: HL237 tablet
- Placebo (Placebo Comparator): Placebo of HL237 tab.
  Interventions: Drug: Placebo of HL237 tablet

INTERVENTIONS:
Drug: HL237 tablet — Treatment A : HL237 100mg, twice a day, Treatment B : HL237 200mg, twice a day, Treatment C : HL237 400mg, twice a day
  Arms: Treatment A; Treatment B; Treatment C
Drug: Placebo of HL237 tablet — Placebo of HL237, twice a day
  Arms: Placebo

SUMMARY:
The purpose of this clinical trial is to determine the optimal dose of HL237 tablets in rheumatoid arthritis patients by comparing the efficacy and safety of the three dose groups of HL237 tablets and the control group.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female, 19 years ≤ age ≤ 80 years
* In the case of women of childbearing age, those who have a negative pregnancy test before randomization
* Patients who agree to use a medically accepted method of contraception during the clinical trial
* Patients corresponding to ACR functional class Ⅰ,Ⅱ,Ⅲ
* Patients with active rheumatoid arthritis with DAS28-ESR > 3.2 in the evaluation of DAS28-ESR identified at the screening
* Patients who were diagnosed with rheumatoid arthritis according to the 2010 ACR/EULAR classification criteria at least 3 months prior to the screening, and showed insufficient response or refractory to treatment with one or more DMARDs.
* Among the subjects who have previously been continuously administering the following rheumatoid arthritis drugs without stopping, those who have used them according to the conditions before randomization and can maintain the current administration regimen and dose during the clinical trial.

  * cDMARDs : Patients who received the same cDMARDs for 12 weeks or more continuously and did not change the dosage and administration of the cDMARDs for 4 weeks or more until the 2nd visit(ex. methotrexate, sulfasalazine, hydroxychloroquine, leflunomide, bucillamine etc.)
  * Prednisolone : Patients who received corticosteroids with a daily dose of 10mg or less of oral prednisolone equivalent continuously, and did not change the dosage and administration for more than 2 weeks until the 2nd visit.
  * Tramadol or NSAIDs : Patients who did not change the dosage and administration for more than 2 weeks consecutively until the 2nd visit
* Patients who have completed the wash-out period as follows until the 2nd visit including the screening period (each period refers to the case where it continues consecutively, and these drugs are contraindicated from the screening).

  * bDMARDs abatacept, adalimumab, certolizumab pegol, golimumab : 10 weeks or more anakinra : 10 days or more etanercept : 3 weeks or more infliximab : 8 weeks or more tocilizumab : 5 weeks or more rituximab : 6 months or more
  * JAK inhibitors tofacitinib, baricitinib : 2 weeks or more
  * immunosuppressants tacrolimus, cyclosporin, azathioprine, cyclophosphamide mizoribine etc : 4 weeks or more
  * tramadol, analgesics and anti-inflammatory analgesic other than NSAIDs : 4 days or more
* Volunteer, be willing and able to provide written informed consent for the trial
* Patients who can read and understand written instructions

Exclusion Criteria:

* Patients corresponding to ACR functional class Ⅳ
* Patients with acquired immune deficiency syndrome or autoimmune diseases other than rheumatoid arthritis
* Severe heart failure, congestive heart failure (NYHA II～IV), ischemic heart disease, peripheral artery disease and/or cerebrovascular disease
* Patients with a history of gastrointestinal bleeding or perforation due to treatment of nonsteroidal anti-inflammatory drugs
* Patients with bleeding or a current history of blood coagulation disorder
* Patients suffering from infectious disease (including tuberculosis, shingles, etc.) at the time of screening or undergoing treatment with the medical history
* Patients with a history of malignant tumors within 5 years prior to screening
* Patients with peptic ulcer confirmed by endoscopy or radiographic examination within 6 months prior to screening
* Patients with a history of gastric or duodenal perforation or obstruction, patients with a history of gastrointestinal surgery (except appendicitis), and patients with a history of upper or lower gastrointestinal bleeding (excluding simple hemorrhoids) within the past year
* Patients with symptoms or signs of pyloric obstruction
* Patients diagnosed with malabsorption within 12 weeks prior to the screening
* Patients with hypersensitive reaction or history of clinically significant hypersensitive reaction to investigational product or its excipients
* Patients with aspirin asthma (asthma attacks caused by nonsteroidal anti-inflammatory drugs) or a history of the same
* Patients with inflammatory bowel disease such as crohn's disease or ulcerative colitis
* Pregnant or breast-feeding
* Patients administered intraarticular, intramuscular, intravenous corticosteroids within 4 weeks priro to the screening.
* Patients with significant psychiatric disorders or taking antidepressants, anticonvulsants, or sedatives
* Patients with substance or alcohol abuse or dependence
* Patients who participate in other clinical trials within 12 weeks prior to the screening and administer investigational drugs or apply clinical trial medical devices
* Patients expected to inevitably administer contraindicated drugs during the clinical trial
* Patients with severe renal dysfuntion(seurum creatinine is 2.0 times higher than the upper limit of normal (based on the institution))
* Patients with severe liver dysfuntion(ALT, AST or total bilirubin is 2.0 times higher than the upper limit of normal (based on the institution))
* Patients that the investigator deems unsuitable for participation in the clinical trial

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2020-09-10 (Actual); Primary Completion 2021-05 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
ACR20(american college of rheumatology 20) response rate | at 12 weeks after administering investigational products
  ACR20(american college of rheumatology 20) response rate at 12 weeks after administering investigational products

SECONDARY OUTCOMES:
ACR20(american college of rheumatology 20) response rate | at 4, 8 weeks after administering investigational products
  ACR20(american college of rheumatology 20) response rate at 4, 8 weeks after administering investigational products
DAS28-ESR(Disease Activity Score 28- erythrocyte sedimentation rate) score | at 4, 8, 12 weeks after administering investigational products
  Change of DAS28-ESR(Disease Activity Score 28- erythrocyte sedimentation rate) score
DAS28-CRP(Disease Activity Score 28-C-reactive protein) score | at 4, 8, 12 weeks after administering investigational products
  Change of DAS28-CRP(Disease Activity Score 28-C-reactive protein) score Change of DAS28-ESR(Disease Activity Score 28- erythrocyte sedimentation rate) score
Tender joint count | at 4, 8, 12 weeks after administering investigational products
  Change of Tender joint count
Swollen joint count | at 4, 8, 12 weeks after administering investigational products
  Change of Swollen joint count
Investigator's composite assessment of disease activity | at 4, 8, 12 weeks after administering investigational products
  Change of Investigator's composite assessment of disease activity (100 mm visual analog scale (0: not active at all, 100: most severely active))
Subject's composite assessment of disease activity | at 4, 8, 12 weeks after administering investigational products
  Change of Subject's composite assessment of disease activity (100 mm visual analog scale (0: not active at all, 100: most severely active))
Subject's assessment of pain (visual analog scale) | at 4, 8, 12 weeks after administering investigational products
  Change of Subject's assessment of pain (100 mm visual analog scale(0: no pain, 100: severe pain))
Subject's assessment of physical function (Korean health assessment questionnaire) | at 4, 8, 12 weeks after administering investigational products
  Change of Subject's assessment of physical function (Korean health assessment
Erythrocyte Sedimentation Rate (ESR) | at 4, 8, 12 weeks after administering investigational products
  Change of Erythrocyte Sedimentation Rate (ESR)
C-Reactive Protein (CRP) | at 4, 8, 12 weeks after administering investigational products
  Change of C-Reactive Protein (CRP)
morning stiffness duration | at 4, 8, 12 weeks after administering investigational products
  Change of morning stiffness duration
The average number of times of use the remedy per day | at 4, 8, 12 weeks after administering investigational products
  Change of The average number of times of use the remedy per day
The percentage of subjects who use the remedy | at 4, 8, 12 weeks after administering investigational products
  Change of the percentage of subjects who use the remedy

CONTACTS AND LOCATIONS:
Locations (1):
- The Catholic University of Korea Seoul ST.MARY'S Hospital, Seoul, South Korea